CLINICAL TRIAL: NCT07024290
Title: Cardiorespiratory Adaptations to High-Intensity Inter-val Training in Young Boxers: A Randomized Con-trolled Study
Brief Title: Cardiorespiratory Adaptations to High-Intensity Inter-val Training in Young Boxers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Collaborators: Kocaeli University (Other)
Responsible Party: Principal Investigator, Monira Aldhahi, Associate prof, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNU-3
Record Dates: First submitted 2025-06-05; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteer; Young
Keywords: high-intensity interval training

STUDY DESIGN:
Intervention Model Description: The experimental group completed a 4-week HIIT-boxing protocol, in addition to regular boxing sessions. HIIT consisted of three weekly sessions, each including three blocks of five 30-second all-out punching intervals on a heavy bag, with 6-second rest between efforts and 1-minute rest between blocks. Heart rate was monitored throughout, confirming training intensities of 88-92% HRmax, consistent with high-intensity training standards in combat sports.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): HIIT consisted of three weekly sessions, each including three blocks of five 30-second all-out punching intervals on a heavy bag, with 6-second rest between efforts and 1-minute rest between blocks.
  Interventions: Behavioral: HITT
- control group (Active Comparator): Participants in both the experimental and control groups followed an identical boxing training program for a period of four weeks, with sessions conducted three times per week. Each session lasted 90 min and was structured in alignment with the established training principles for amateur boxing. The training began with a 15-minute general warm-up phase, including dynamic mobility drills and calisthenics, to elevate core temperature and enhance neuromuscular readiness.
  Interventions: Other: Regular training

INTERVENTIONS:
Behavioral: HITT — The experimental group completed a 4-week HIIT-boxing protocol, in addition to regular boxing sessions. HIIT consisted of three weekly sessions, each including three blocks of five 30-second all-out punching intervals on a heavy bag, with 6-second rest between efforts and 1-minute rest between blocks. Heart rate was monitored throughout, confirming training intensities of 88-92% HRmax, consistent with high-intensity training standards in combat sports.
  Arms: Exercise group
Other: Regular training — Participants in control groups followed a boxing training program for a period of four weeks, with sessions conducted three times per week. Each session lasted 90 min and was structured in alignment with the established training principles for amateur boxing. The training began with a 15-minute general warm-up phase, including dynamic mobility drills and calisthenics, to elevate core temperature and enhance neuromuscular readiness.
  Arms: control group

SUMMARY:
This study examined the effects of a structured 4-week high-intensity interval training (HIIT) program integrated with boxing on young trained individuals. Participants were randomly assigned to a HIIT-boxing group or a control group. Pre- and post-intervention assessments measured pulmonary function, aerobic capacity (VO₂max), and heart rate recovery (HRR) at 1, 3, and 5 minutes post-exercise. The study aimed to explore physiological adaptations, particularly improvements in cardiopulmonary and autonomic function.

Integrating HIIT with boxing training may serve as an effective conditioning strategy for enhancing aerobic fitness, pulmonary function, and autonomic cardiovascular regulation in trained individuals. This combined approach could be valuable in sports performance programs and rehabilitation settings where improving VO₂max and recovery efficiency is a priority.

DETAILED DESCRIPTION:
Background: High-intensity interval training (HIIT) has been recognized for its effectiveness in enhancing cardiorespiratory fitness. However, their combined application in boxing training remains underexplored. This study aimed to investigate the physiological adaptations induced by a structured 4-week HIIT-boxing regimen, with a specific focus on pulmonary function, aerobic capacity, and autonomic cardiovascular regulation, assessed by heart rate recovery (HRR). Methods: Sixteen trained young individuals were randomly assigned to either the HIIT-boxing group or the control group. Comprehensive assessments, including pulmonary function tests, peak oxygen uptake (VO2max), and HRR at the 1st, 3rd, and 5th minutes post-exercise, were conducted pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-30 years.
* Actively engaged in structured boxing training for at least 2 years.
* Training a minimum of 3 days per week.
* Free of cardiovascular, pulmonary, or neuromuscular conditions.
* Willing to abstain from non-study physical training 48 hours prior to testing.
* Provided written informed consent after receiving a full explanation of study procedures.

Exclusion Criteria:

* Had any diagnosed medical conditions contraindicating high-intensity exercise (e.g., uncontrolled asthma, cardiac arrhythmias).
* Reported current musculoskeletal injuries limiting full participation.
* Were taking medications affecting heart rate or respiratory function.
* Missed more than 10% of the assigned training sessions.
* Failed to adhere to pre-assessment instructions (e.g., rest or diet restrictions).

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | baseline and after 4 weeks
  Pulmonary function tests were performed using a calibrated desktop spirometer (COSMED Pony FX; COSMED, Rome, Italy) to assess the key respiratory parameters. FVC was recorded to assess lung volume and respiratory strength. Participants performed a maximal inhalation followed by a forceful exhalation to expel as much air as possible.
  Unit of Measure: Liters (L)
Aerobic Capacity | baseline and after 4 weeks
  Aerobic capacity was determined using the Yo-Yo Intermittent Recovery Level 1 (Yo-Yo IR1) test, a validated method for assessing maximal aerobic capacity in intermittent sports. The participants completed repeated 20-meter shuttle runs at increasing speeds, with short recovery periods between efforts. The aerobic capacity was predicted using the established regression equations for the Yo-Yo IR1 test.
Maximal Voluntary Ventilation (MVV) | Baseline and after 4 weeks
  MVV was measured using a calibrated desktop spirometer (COSMED Pony FX; COSMED, Rome, Italy) to evaluate overall ventilatory capacity. Participants were instructed to breathe in and out as rapidly and deeply as possible for 12-15 seconds; the value was extrapolated to represent the maximum volume of air inhaled and exhaled in one minute (L/min).
  Unit of Measure: Liters per minute (L/min)
Forced Expiratory Volume in One Second (FEV1) | Baseline and after 4 weeks
  FEV1 was measured as the volume of air forcefully exhaled in the first second of the FVC maneuver. This value reflects airway patency and expiratory power.
  Unit of Measure: Liters (L)
Peak Expiratory Flow (PEF) | Baseline and after 4 weeks
  PEF was assessed to determine the highest speed at which air can be expelled from the lungs during a forceful exhalation following full inspiration.
  Unit of Measure: Liters per minute (L/min)

CONTACTS AND LOCATIONS:
Overall Officials: Cinarli, Principal Investigator — Department of Physiotherapy and Rehabilitation, Kocaeli Health and Technology University, Kocaeli,
Locations (1):
- Sena Cinarli, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided